CLINICAL TRIAL: NCT04645433
Title: Effect of Favipiravir on Mortality in Patients With COVID-19 at a Tertiary Center Intensive Care Unit: Single Center Experience
Brief Title: Effect of Favipiravir on Mortality in Patients With COVID-19 at a Tertiary Center Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sultan Acar Sevinç, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2854
Record Dates: First submitted 2020-11-07; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Mortality; Intensive Care Unit
Keywords: covid 19; favipiravir
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Favipiravir therapy: Favipiravir was advised to all patients with severe pneumonia and progressing pneumonia findings or worsening clinical manifestations except pregnant, breast feeding, postpartum woman. PCR results were not waited to start favipiravir in this group of patients and continued if it would be negative but tomography findings were consistent with COVID-19. Loading dose was 1600 mg twice a day. Maintenance dose was 600 mg per 12 hours for four days.
- Lopinavir-ritonavir therapy: Lopinavir-ritonavir therapy was used in selected ICU patients before widespread availability of favipiravir (23 March 2020) and/or if favipiravir was contraindicated. Combination of lopinavir 200 mg-ritonavir 50 mg tablet was the given form. It was given as double tablets twice daily for 10-14 days. Patients were accepted as under favipiravir therapy if they had incomplete course of lopinavir-ritonavir therapy (less than 5 days) and followed by favipiravir for 5 days.

SUMMARY:
Effect of Favipiravir and Lopinavir-Ritonavir on Mortality in a Tertiary Center Intensive Care Unit: Single Center Experience

DETAILED DESCRIPTION:
Many agents have been given for treatment of COVID-19 infection. "Covid-19 Diagnosis and Treatment Guideline" by Ministry of Health was advised nationwide use of favipiravir or lopinavir-ritonavir although evidence was scarce for the nationwide use of lopinavir-ritonavir or favipiravir to treat COVID-19 at the time of publication date of detailed guideline Favipiravir is a RNA dependent RNA polymerase inhibitor and approved for treatment of influenza in Japan at 2014 The aim of the study was to compare ICU and hospital mortality in patients with favipiravir or lopinavir-ritonavir treatment and compare other laboratory parameters in patients treated with these two antiviral agents.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older

Exclusion Criteria:

* patients younger than 18 years old
* patients who have received both lopinavir-ritonavir and favipiravir sepuentially

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care units (ICU) between March o 10thand May 10th 2020 due to COVID-19 infection were included to the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality for ICU | 14 days
  If the patient dies, we have reached an outcome
hospital stay | 14 days
  If the hospital stay exceeds 14 days, we have reached an outcome

CONTACTS AND LOCATIONS:
Overall Officials: sultan acar sevinc, Principal Investigator — Sisli Hamidiye Etfal Education and Training Hospital
Locations (1):
- SisliHamidiye Etfal Education and Training Hospital, Istanbul, Turkey (Türkiye)